CLINICAL TRIAL: NCT00413569
Title: The Effect of Intubation Method on Outcome of Cervical Spine Surgery
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Other Study IDs: 0610008805
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Last update posted 2006-12-19 (Estimated); Status verified 2006-12

CONDITIONS: Cervical Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

INTERVENTIONS:
Procedure: cervical spine surgery

SUMMARY:
The specific aim of this study is to demonstrate that inserting a breathing tube using a standard laryngoscope with the patient fully anesthetized is a safe and effective means of securing the airway in a patient with cervical spine disk herniation or stenosis. The two groups compared are composed of those who are intubated with direct laryngoscopy and those who are intubated with a fiberoptic scope.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age for cervical disk herniation or cervical spine surgery by either Drs Snow or Lavyne from 1998-2006.

Exclusion Criteria:

* Unstable (broken) cervical spine

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Solomon, MD, Principal Investigator — Weill Medical College of Cornell University